CLINICAL TRIAL: NCT04877522
Title: An Open Label, Multi-center Asciminib Roll-over Study to Assess Long-term Safety in Patients Who Have Completed a Novartis Sponsored Asciminib Study and Are Judged by the Investigator to Benefit From Continued Treatment
Brief Title: Asciminib Roll-over Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CABL001A2001B; 2021-000602-17 (EudraCT Number); 2023-507557-16-00 (Other: EU CTIS)
Expanded Access: NCT04360005 (Available)
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Chronic Myelogenous Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive
Keywords: Chronic Myelogenous Leukemia; CML; ALL; CML-AP; CML-BP; CML-CP; myeloproliferative neoplasm; chronic phase; accelerated phase; blast phase; ABL001; asciminib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myeloproliferative Disorders; Blast Crisis | interventions — asciminib; Imatinib Mesylate; nilotinib; bosutinib; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Asciminib single agent group (Experimental): Participants with CML or ALL, from Novartis sponsored asciminib studies, including but not limited to CABL001A2301, CABL001A2302, CABL001X2101, CABL001A2202, CABL001AUS04 and CABL001AUS08 studies, that were receiving asciminib
  Interventions: Drug: Asciminib single agent
- Bosutinib single agent group (Other): Participants with CML-CP, from Novartis sponsored asciminib study CABL001A2301, that were receiving bosutinib
  Interventions: Drug: Bosutinib
- Bosutinib-Asciminib switch group (Experimental): Participants with CML-CP, from Novartis sponsored asciminib study CABL001A2301 that were receiving bosutinib treatment and switched to asciminib when entering this study or during the course of this study
  Interventions: Drug: Asciminib single agent
- Asciminib in combination with imatinib group (Experimental): Participants with CML from Novartis sponsored asciminib studies CABL001E2201 or CABL001X2101 that were receiving asciminib combined with imatinib
  Interventions: Drug: Imatinib
- Asciminib in combination with nilotinib group (Experimental): Participants with CML or ALL from Novartis sponsored asciminib studies CABL001E2201or CABL001X2101 that were receiving asciminib combined with nilotinib
  Interventions: Drug: Nilotinib
- Imatinib single agent group (Other): Participants with CML-CP, from Novartis sponsored asciminib study CABL001E2201 that were receiving imatinib
  Interventions: Drug: Imatinib
- Nilotinib single agent group (Other): Participants with CML-CP, from Novartis sponsored asciminib study CABL001E2201 and CABL001J12302 that were receiving nilotinib
  Interventions: Drug: Nilotinib
- Asciminib in combination with dasatinib group (Experimental): Participants with CML from Novartis sponsored study CABL001X2101 that were receiving asciminib with dasatinib
  Interventions: Drug: Dasatinib
- Dasatinib single agent group (Other): Participant with CML-CP , from Novartis sponsored asciminib study CABL001A2202, CABL001J12301, that were receiving Dasatinib.
  Interventions: Drug: Dasatinib
- Dasatinib-Asciminib switch group (Experimental): Participants with CML-CP, from Novartis sponsored asciminib study CABL001A2202 that were receiving best available therapy (dasatinib) and switched to asciminib when entering this study or during the course of this study
  Interventions: Drug: Asciminib single agent
- Asciminib single agent formulation for Pediatric (Experimental): Participants with CML, from Novartis sponsored asciminib studies, including but not limited to CABL001I12201 study, that were receiving asciminib
  Interventions: Drug: Asciminib single agent pediatric formulation

INTERVENTIONS:
Drug: Asciminib single agent — Taken orally, twice daily (BID) or once daily (QD), in fasting state
  Other Names: ABL001
  Arms: Asciminib single agent group; Bosutinib-Asciminib switch group; Dasatinib-Asciminib switch group
Drug: Imatinib — Taken orally, once daily, in the morning with low-fat meal
  Other Names: STI571
  Arms: Asciminib in combination with imatinib group; Imatinib single agent group
Drug: Nilotinib — Taken orally, twice daily, on an empty stomach
  Other Names: AMN107
  Arms: Asciminib in combination with nilotinib group; Nilotinib single agent group
Drug: Bosutinib — Taken orally, once daily, with food
  Arms: Bosutinib single agent group
Drug: Dasatinib — Taken orally, once daily in a fasted state, 1 or 2 hours before a meal
  Other Names: Sprycel
  Arms: Asciminib in combination with dasatinib group; Dasatinib single agent group
Drug: Asciminib single agent pediatric formulation — Pediatric participants receive a body weight adjusted dose of 1.3 mg/kg of pediatric film coated granules with food twice daily (b.i.d.) or 2.6 mg/kg once daily (q.d.) in the morning.
  Other Names: ABL001
  Arms: Asciminib single agent formulation for Pediatric

SUMMARY:
This is a long term safety study for patients who have completed a Novartis sponsored asciminib study and are judged by the investigator to benefit from continued treatment

DETAILED DESCRIPTION:
This is an open-label, multi-center, global roll-over study designed to assess long term safety and provide continued treatment to participants who have previously participated in an asciminib Novartis sponsored study and who, in the opinion of the investigator, would benefit from continued treatment as in their parent study but are unable to access this treatment outside of the clinical study.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participant with PH+ CML or PH+ ALL currently receiving treatment with asciminib (single agent or in combination with imatinib, nilotinib or dasatinib), imatinib, nilotinib or bosutinib alone within a Novartis-sponsored study and, in the opinion of the Investigator, would benefit from continued treatment.
2. Participant has demonstrated compliance on the parent study protocol and is willing and able to comply with scheduled visits, treatment plans and any other study procedures.

Key Exclusion Criteria:

1. Participant has been discontinued from parent study treatment.
2. Participant currently has unresolved toxicities reported as possibly related to study treatment in the parent study.
3. Participant's ongoing treatment is currently approved and reimbursed at country level.
4. Pregnant or nursing (lactating) women.
5. Women of child-bearing potential, unless they are using highly effective methods of contraception and willing to continue while taking study treatment.
6. Sexually active males receiving imatinib, nilotinib, bosutinib or dasatinib unwilling to follow the relevant contraception requirements in the local prescribing information.
7. Applicable for participants on bosutinib treatment at the end of the CABL001A2301 and on other TKIs for CABL001A2202 study that switch to asciminib treatment:

   * Asymptomatic (grade 2) pancreatitis if not resolved within 28 days
   * QTcF>480msec or inability to determine QTc interval
   * any grade 3 or 4 toxicity not resolved to grade 2 or lower within 28 days before starting asciminib treatment

Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 7 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 347 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2030-08-29 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | 8 years
  All AEs and SAEs will be tabulated and listed for participants in the Safety Set by treatment group. From day of first administration of study treatment to 30 days after the last study treatment.

SECONDARY OUTCOMES:
Percentage of participants with clinical benefit as assessed by Investigator | 8 years
  Investigators' assessment of clinical benefit will collected through the Investigator confirming that the patient is still benefiting from treatment. This will be evaluated and tabulated for participants in the Safety Set by treatment group at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (77):
- United States (5):
  - Michigan Med University of Michigan, Ann Arbor, Michigan
  - Memorial Sloan Kettering, New York, New York
  - Oregon Health Sciences University, Portland, Oregon
  - Texas Oncology, Dallas, Texas
  - Uni Of TX MD Anderson Cancer Cntr, Houston, Texas
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Capital Federal
- Austria (2):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Vienna
- Brazil (2):
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Varna, Bulgaria
- Novartis Investigative Site, Montreal, Quebec, Canada
- China (11):
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Shenyang
  - Novartis Investigative Site, Tianjin
- Czechia (2):
  - Novartis Investigative Site, Ostrava, Poruba
  - Novartis Investigative Site, Brno
- Novartis Investigative Site, Copenhagen, Denmark
- France (6):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (4):
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Kiel
- Italy (3):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Kobe, Japan
- Novartis Investigative Site, Beirut, Lebanon
- Malaysia (3):
  - Novartis Investigative Site, George Town, Pulau Pinang
  - Novartis Investigative Site, Johor Bahru
  - Novartis Investigative Site, Kuala Selangor
- Novartis Investigative Site, Monterrey, Nuevo León, Mexico
- Novartis Investigative Site, Khoudh, Oman
- Poland (4):
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Portugal (2):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Novartis Investigative Site, Timișoara, Romania
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Singapore, Singapore
- South Korea (4):
  - Novartis Investigative Site, Uijeongbu-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Jeollanam
- Spain (9):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Badalona, Barcelona
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Bilbao, Bizkaia
  - Novartis Investigative Site, Santa Cruz, Santa Cruz De Tenerife
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Novartis Investigative Site, Taoyuan District, Taiwan
- Novartis Investigative Site, Samsun, Atakum, Turkey (Türkiye)
- United Kingdom (2):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Oxford
- Vietnam (2):
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
Supporting Information: CSR